CLINICAL TRIAL: NCT01611805
Title: A Placebo-Controlled, Four-Period Crossover, Single Ascending Oral Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of the CCR9 Receptor Antagonist GSK1605786 in Japanese Healthy Male Subject
Brief Title: Japanese Phase I of GSK1605786
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 114472
Record Dates: First submitted 2012-04-12; First posted 2012-06-05 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- GSK1605786 250mg (Experimental): Opaque Swedish orange body and cap.
  Interventions: Drug: GSK1605786
- Placebo (Placebo Comparator): Opaque Swedish orange body and cap.
  Interventions: Drug: GSK1605786 Placebo
- GSK1605786 500mg (Experimental): Opaque Swedish orange body and cap.
  Interventions: Drug: GSK1605786
- GSK1605786 1000mg (Experimental): Opaque Swedish orange body and cap.
  Interventions: Drug: GSK1605786
- GSK1605786 500mg in fed (Experimental): Opaque Swedish orange body and cap.
  Interventions: Drug: GSK1605786

INTERVENTIONS:
Drug: GSK1605786 — Opaque Swedish orange body and cap.
  Arms: GSK1605786 1000mg; GSK1605786 250mg; GSK1605786 500mg; GSK1605786 500mg in fed
Drug: GSK1605786 Placebo — Opaque Swedish orange body and cap.
  Arms: Placebo

SUMMARY:
This is an double-blind, single dose, four-period, crossover study in Japanese healthy male volunteers to assess the pharmacokinetics and safety/tolerability of single doses of GSK1605786A. Approximately 24 subjects will receive three treatments of 250, 500, and 1000mg GSK1605786 under fasted conditions or 500mg after food intake plus placebo in a dose ascending crossover design. Serial pharmacokinetic samples will be collected following each dose and safety assessments will be performed. The pharmacokinetics and dose proportionality of GSK1605786 after single oral doses of GSK1605786 at the dose levels of 250mg, 500mg and 1000 mg under fasted conditions will be assessed. In addition, a comparison will be made between the pharmacokinetics of GSK1605786 under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese as
* Japanese defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity -Male between 20 and 55 years of age inclusive, at the time of signing the informed consent.
* Body weight =>50kg and BMI within the range 18.5 - 25 kg/m2 (inclusive).

Exclusion Criteria:

- Known coeliac disease or positive serologic testing for anti-tTG antibodies (required to screen for undiagnosed celiac disease)

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07-22 (Actual); Primary Completion 2010-10-06 (Actual); Study Completion 2010-10-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentration | up to 72h post dose

SECONDARY OUTCOMES:
Adverse envents | up to 72h post dose
Vital signe | up to 72h post dose
Clinical laboratory | up to 72h post dose
12 lead ECG | up to 72h post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

REFERENCES:
- See also: Results for study 114472 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114472?search=study&search_terms=114472#rs